CLINICAL TRIAL: NCT00725491
Title: A Phase III, Multi-center, Open-label, Randomized Study to Assess the Efficacy and Safety of Org 37462 Treatment in Chinese Women Undergoing Controlled Ovarian Stimulation for IVF or ICSI, Using a Long Protocol of Triptorelin as a Reference Treatment.
Brief Title: A Study to Assess the Efficacy and Safety of Ganirelix (Orgalutran®) Treatment in Chinese Women Undergoing Controlled Ovarian Stimulation for in Vitro Fertilization (IVF) or Intra Cytoplasmatic Sperm Injection (ICSI) (Study 38651)(P05703)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P05703; 38651
Record Dates: First submitted 2008-07-28; First posted 2008-07-30 (Estimated); Results first posted 2010-01-22 (Estimated); Last update posted 2022-02-03 (Actual); Status verified 2022-02

CONDITIONS: Controlled Ovarian Stimulation
Keywords: Reproductive; techniques; assisted
MeSH Terms: conditions — Helping Behavior | interventions — ganirelix; Triptorelin Pamoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): ganirelix
  Interventions: Drug: ganirelix
- 2 (Active Comparator): triptorelin
  Interventions: Drug: triptorelin

INTERVENTIONS:
Drug: ganirelix — On day 6 of recFSH treatment, Org 37462 treatment will start by daily SC administration (0.25 mg) up to and including the day of hCG administration.
  Other Names: Orgalutran®; Org 37462
  Arms: 1
Drug: triptorelin — a daily dose of 0.05 mg SC is to be injected. Triptorelin treatment will start in the luteal phase at day 21-24 of the menstrual cycle. Treatment with recFSH will start 14 days later if treatment with triptorelin has resulted in downregulation, i.e. serum E2 <= 50 pg/ml (<= 200pmol/l). In case the hypogonadotropic state is not reached after 14 days of pretreatment, the dose of triptorelin will be increased to 0.1 mg. If downregulation is not reached within 28 days of pre-treatment with triptorelin, the subject will be discontinued from further hormonal treatment. The daily dose of triptorelin is sustained up to and including the day of hCG.
  Other Names: Decapeptyl
  Arms: 2

SUMMARY:
The primary purpose of this study is to assess that ganirelix is safe and well-tolerated in Chinese women and that a controlled ovarian stimulation (COS) protocol combining recombinant follicle stimulating hormone (recFSH) with ganirelix is efficient in Chinese women undergoing COS for in vitro fertilization (IVF) or intra cytoplasmatic sperm injection (ICSI).

ELIGIBILITY:
Inclusion Criteria:

* females of infertile couples for whom COS and IVF or ICSI is indicated
* body mass index between 18 and 29 kg/m2
* willing and able to give written informed consent.

Exclusion Criteria:

* More than three previous COS cycles for assisted reproduction since last established ongoing pregnancy (if applicable)
* History of no or low ovarian response to FSH/human menopausal gonadotropin (hMG) treatment
* Less than 2 ovaries or any other ovarian abnormality including endometrioma
* Presence of unilateral or bilateral hydrosalpinx
* Any ovarian and/or abdominal abnormality that would interfere with adequate ultrasound investigation of at least one ovary
* History of or current polycystic ovary syndrome (PCOS)
* History of/or current endocrine abnormality
* Any clinically relevant hormone value outside the reference range during the early follicular phase
* Any clinically significant abnormal laboratory value
* Hypertension or currently treated hypertension
* Recent history of current epilepsy, diabetes, cardiovascular, gastro-intestinal, hepatic, renal, pulmonary disease
* Alcohol or drug abuse, or history thereof
* Current serious allergic symptoms
* Abnormal cervical smear
* Known hypersensitivity to gonadotropin releasing hormone (GnRH) or its analogs;
* Contra-indications for the use of gonadotropins
* Use of hormonal preparations within 1 month prior to the date of signing consent;
* Administration of any investigational product within 3 months prior to screening.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 259 (Actual)
Dates: Start 2007-05; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

REFERENCES:
- [Derived] Qiao J, Lu G, Zhang HW, Chen H, Ma C, Olofsson JI, Witjes H, Heijnen E, Mannaerts B. A randomized controlled trial of the GnRH antagonist ganirelix in Chinese normal responders: high efficacy and pregnancy rates. Gynecol Endocrinol. 2012 Oct;28(10):800-4. doi: 10.3109/09513590.2012.665103. Epub 2012 Mar 20. PMID 22429192

RESULTS

PARTICIPANT FLOW:
Groups:
- Ganirelix: 0.25 mg once daily from stimulation day 6 onwards up to the day of human chorionic gonadotropin (hCG).
- Triptorelin: 0.05 mg once daily from cycle day 21-24 onwards up to the day of hCG
Period: Overall Study
Arm/Group | Ganirelix | Triptorelin
Started | 113 (Intent-to-Treat Group) | 120 (Intent-to-Treat Group)
Completed | 104 | 102
Not Completed | 9 | 18
Not completed — Adverse Event | 3 | 2
Not completed — Pregnancy | 0 | 3
Not completed — Risk for hyperstimulation | 2 | 9
Not completed — No/too few oocytes/bad quality oocytes | 1 | 1
Not completed — Fertilization failure | 0 | 1
Not completed — No/too few embryos/ bad quality embryos | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ganirelix | Triptorelin | Total
Number analyzed (Participants) | 113 | 120 | 233
Age, Continuous [Mean (Standard Deviation); unit: years] — Intention to treat population
  years | 29.3 (2.8) | 29.1 (3.0) | 29.2 (2.9)
Sex: Female, Male [Count of Participants; unit: Participants] — Intention to treat population
  Participants
    Female | 113 | 120 | 233
    Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — Intention to treat population
  participants
    China | 113 | 120 | 233

OUTCOME MEASURES:

1. Primary Outcome: The Amount of International Units (IU) of Recombinant Follicle Stimulating Hormone (recFSH) Needed in a Controlled Ovarian Stimulation (COS) Cycle up to the First Day the Human Chorionic Gonadotropin (hCG) Criterion is Met.
Description: The hCG criterion is met the first day that 3 follicles >= 17 mm are observed.
Time Frame: At completion of ovarian stimulation; maximally after 18 days of recFSH administration.
Population: The number of participants for this analysis included only those participants in the intent-to-treat (ITT) group who received hCG and for whom data was available.
Measure: Mean (Standard Deviation); unit: international units (IU)
Arm/Group | Ganirelix | Triptorelin
Number analyzed (Participants) | 109 | 114
international units (IU) | 1272.0 (265.8) | 1415.6 (355.6)
Statistical Analysis 1: Comparison: Ganirelix vs Triptorelin; Test type: Superiority or Other; p < 0.001, Cochran-Whitehead

ADVERSE EVENTS:
Description: One subject in the ganirelix group started ovarian stimulation with recFSH but was never treated with ganirelix.
Arm/Group | Ganirelix | Triptorelin
Serious Adverse Events (participants affected / at risk) | 4/112 | 2/120
Other Adverse Events (participants affected / at risk) | 13/112 | 13/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ganirelix (N=112) | Triptorelin (N=120)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0)
Ovarian hyperstimulation syndrome (Reproductive system and breast disorders) | 1 (1) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ganirelix (N=112) | Triptorelin (N=120)
Nausea (Gastrointestinal disorders) | 9 (9) | 11 (11)
Vomiting (Gastrointestinal disorders) | 6 (6) | 7 (7)
Antepartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 6 (6) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review any scientific paper, presentation, or other communication concerning the clinical trial at least 6 weeks ahead of estimated publication or presentation. In order to protect its proprietary interests, the sponsor shall have the right to make its consent, which shall not be withheld unreasonably, conditional upon proper representation of the interpretation of both the sponsor and the investigator(s) in the discussion of the data in such communications.